CLINICAL TRIAL: NCT04789096
Title: A Phase II, Two-arm, Non-comparative, Multicentre Study of Tucatinib (ONT-380), Pembrolizumab and Trastuzumab in Patients With Pre-treated Advanced HER2-positive Breast Cancer
Brief Title: Tucatinib Together With Pembrolizumab and Trastuzumab
Acronym: TUGETHER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped on the recommendation of the BCT Independent Data and Monitoring Committee
Sponsor: Breast Cancer Trials, Australia and New Zealand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCT 2102
Record Dates: First submitted 2021-03-01; First posted 2021-03-09 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tucatinib; pembrolizumab; Trastuzumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TUGETHER Treatment (Experimental): Participants will receive:
  * Tucatinib (oral) at a dose of 300 mg BD on day 1-21 of each 21-day cycle
  * Pembrolizumab will be administered at a dose of 200 mg IV on day 1 of each 21 day cycle
  * Trastuzumab will be given as a loading dose of 8 mg/kg IV (if loading required, otherwise 6 mg/kg) on day 1 followed by 6 mg/kg on day 1 of each 21 day cycle.
  Participants registered to PD-L1 negative/unknown cohort prior to Protocol Amendment 2 received Capecitabine 1000 mg/m^2 day 1-14 of each 21 day cycle.
  Interventions: Drug: Tucatinib; Drug: Pembrolizumab; Drug: Trastuzumab; Drug: Capecitabine

INTERVENTIONS:
Drug: Tucatinib — Oral tablet
  Other Names: Tukysa
Drug: Pembrolizumab — Intravenous
  Other Names: Keytruda
Drug: Trastuzumab — Intravenous
  Other Names: Herceptin
Drug: Capecitabine — Oral tablet
  Other Names: Xeloda

SUMMARY:
Women or men with HER2-positive, metastatic breast cancer, who have progressed on previous treatment, will receive tucatinib in combination with pembrolizumab and trastuzumab (PD-L1 positive).

DETAILED DESCRIPTION:
Despite significant advances in systemic treatment options, advanced HER2-positive breast cancer post treatment with trastuzumab, pertuzumab and T-DM1 still remains incurable, with brain metastases remaining a major cause of patient morbidity and mortality.

HER2-positive breast cancers have relatively high tumour infiltrating lymphocytes (TILs) that may be targeted with immune checkpoint blockade. Studies in metastatic breast cancer with PD1 or PD-L1 inhibition have shown an overall survival (OS) benefit for those that are enriched for pre-existing immunity, such as positive expression of PD-L1 protein or TILs present.

One of the main areas of disease progression in HER2 positive disease is in the central nervous system (CNS), supporting the need to find an effective combination for patients with brain metastases.

Tucatinib (ONT-380) is a potent, highly selective, oral HER2 small molecule tyrosine kinase inhibitor (TKI) with demonstrated clinical benefit notable for its minimal inducement of EGFR-type toxicities when administered in combination-type studies including proven intra-cranial efficacy in studies of patients with brain metastases.

The investigators hypothesise that the combination of tucatinib with trastuzumab and PD-1 inhibition will result in a similar ORR as that seen in HER2CLIMB, along with comparable PFS and duration of response, particularly through prevention and treatment of CNS metastases. The potential advantage of adding PD-1 inhibition and omitting capecitabine in the PD-L1 positive group is to increase the durability of the response, with hopefully less added toxicity for patients. The investigators believe this regimen will result in comparable outcomes as those seen in HER2CLIMB, with fewer adverse events. Importantly, the side effect profiles of all agents in our proposed combination are non-overlapping and this combination provides a unique opportunity for excellent tolerability and durable disease control in this patient group. The study design initially included two treatment cohorts, with the PD-L1 negative/unknown cohort being treated with the HER2CLIMB regimen with the addition of pembrolizumab (MK-3475), under the hypothesis that the anti-tumour activity of this regimen will overcome the lower immunogenicity of this subgroup. However, Protocol Amendment 2 will omit capecitabine in the PD-L1 negative/unknown cohort due to a high frequency of liver test abnormalities within the first seven participants in this cohort.

ELIGIBILITY:
Inclusion Criteria (Pre-Registration):

1. Has provided written, informed consent to participate in the study.
2. Female or male, age ≥ 18 years.
3. Local histologically confirmed HER2-positive unresectable loco-regional or metastatic breast cancer. HER2-positive according to ASCO CAP 2018 guidelines defined as:

   1. ISH testing with ERBB2-amplification as demonstrated by ratio ERBB2/centromeres ≥ 2.0 or mean gene copy number ≥ 6 OR
   2. 3+ staining by IHC.
4. FFPE tumour samples (preferably two blocks) available from newly obtained biopsies of advanced disease for assessment of PD-L1, TILs status and correlative research. If new biopsies are not obtainable then primary/metastatic archival biopsies (preferably two samples) from within 12 months of registration may be provided.For those participants whose tissue is unavailable despite best efforts (e.g. inadequate sample or primary tumour lost/discarded), please discuss with BCT and the Study Chairs.
5. Must have previously received taxane, trastuzumab, pertuzumab and an antibody-drug conjugate (ADC) in either the (neo) adjuvant or advanced disease setting. Any number of prior lines of anti-HER2 therapy is acceptable.
6. Have progression of unresectable locally advanced or metastatic breast cancer during or after last systemic therapy (as confirmed by investigator), or be intolerant of last systemic therapy.
7. Have a life expectancy of at least 6 months, in the opinion of the investigator.
8. Women of childbearing potential (WOCBP) and men with partners of childbearing potential must agree to use a highly effective contraception from the signing of informed consent until 7 months after the last dose of protocol treatment.

   Note: Use of oral, injectable or implant hormonal contraceptives or medicated IUD must stop before registration.
9. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations during both the treatment and follow-up phases.

Inclusion Criteria (Registration):

In addition to the above listed pre-registration inclusion criteria, participants must fulfill all the following criteria before registration:

1. Confirmed submission to the central laboratory of tumour tissue for PD-L1 status to determine cohort . For those participants whose tissue is unavailable for testing, individual cases must be discussed with BCT and the Study Chairs. Note: the first 10 participants will be reviewed for PD-L1 positivity rates
2. Have Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
3. Have measurable disease assessable by RECIST v1.1.
4. Must have one of the following (based on screening brain MRI):

   a) No evidence of brain metastases OR b) Untreated brain metastases not needing immediate local therapy. Participants with CNS measurable disease by RECIST 1.1 criteria, with or without measurable extracranial disease by RECIST are eligible. For participants with untreated CNS lesions > 2.0 cm on screening MRI, discussion with and approval from BCT and the Study Chair is required before registration OR c) Previously treated brain metastases: i) Brain metastases previously treated with local therapy may either be stable since treatment or may have progressed since prior local brain metastasis therapy, provided that there is no clinical indication for immediate re-treatment with local therapy in the opinion of the investigator.

   ii) Participants treated with CNS local therapy for newly identified lesions found on initial MRI performed during screening for this study may be eligible if the following criteria are met: (1) Time since whole brain radiation therapy (WBRT) is ≥ 14 days before registration, or (2) Time since stereotactic radiosurgery is ≥ 7 days before registration, or time since surgical resection is ≥ 28 days (3) Other sites of disease assessable by RECIST 1.1. are present.
5. Relevant records of any CNS treatment must be available to allow for classification of target and non-target lesions.
6. Have a left ventricular ejection fraction (LVEF) of ≥ 50% as assessed by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA) documented within 8 weeks before registration.
7. Have adequate haematological, coagulation, hepatic and renal functions within 7 days before registration as defined as:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
   2. Platelet count ≥ 100 x 10^9/L
   3. Haemoglobin ≥ 90 g/L
   4. Creatinine ≤ 1.5 x ULN or serum creatinine clearance > 40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance:
   5. Serum total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). In the case of known Gilbert's disease, serum total bilirubin < 2 x ULN is allowed
   6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x institutional ULN unless liver metastases are present, in which case it must be ≤ 5 x ULN
   7. International normalised ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless on medication known to alter INR and aPTT (Note: Warfarin and other coumarin derivatives are prohibited).
8. Evidence of post-menopausal status, or negative urine or serum pregnancy test for female pre-menopausal participants. Women who have undergone surgical sterilisation (bilateral oophorectomy, bilateral salpingectomy/tubal ligation, or hysterectomy) do not require pregnancy testing. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   1. Women < 50 years of age would be considered post-menopausal/non-fertile if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments or chemotherapy (whichever is most recent) and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution.
   2. b) Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, or had chemotherapy-induced menopause with last menses > 1 year ago.

Exclusion Criteria (Pre-Registration):

Any one of the following is regarded as a criterion for exclusion from pre-registration to the study:

1. Previously treated with:

   1. Lapatinib within 12 months of registration OR
   2. Neratinib or afatinib within 12 months of registration, unless ceased due to toxicity and not progression.
2. Prior anti-PD-1, anti-PD-L1/L2 or anti-CTLA4 therapy, including, but not limited to: pembrolizumab, nivolumab, atezolizumab, durvalumab, avelumab, ipilimumab, tremelimumab.
3. Previous severe hypersensitivity reaction to treatment with TKI or monoclonal antibody that is biologically similar to the study treatments.
4. Known leptomeningeal disease as documented/determined by the investigator.
5. Have poorly controlled (> 1/week) generalised or complex partial seizures, or manifest neurologic progression due to brain metastases despite CNS-directed therapy.
6. History of clinically significant or uncontrolled cardiac disease, including congestive heart failure (New York Heart Association functional classification ≥ 3), angina, myocardial infarction or ventricular arrhythmia. Have known myocardial infarction or unstable angina within 6 months before registration.
7. Active or history of autoimmune disease or immune deficiency, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

   1. History of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible
   2. Stable diabetes mellitus are eligible
   3. Eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g. patients with psoriatic arthritis are excluded) are eligible provided ALL the following conditions are met:

   i) Rash must cover < 10% of body surface area ii) Disease is well controlled at baseline and requires only low-potency topical corticosteroids iii) No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
8. Known human immunodeficiency virus (HIV) (HIV1/2antibodies) or active Hepatitis B (HBsAg reactive) or Hepatitis C (HCV RNA [qualitative]).

   1. Participants with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible
   2. Participants positive for HCV antibody are eligible only if polymerase change reaction is negative for HCV RNA.
9. Pregnant, breastfeeding or planning a pregnancy; lactating participants must stop breast feeding before registration.
10. Require therapy with warfarin or other coumarin derivatives (non-coumarin anticoagulants are allowed).
11. Unable to swallow pills or has significant gastrointestinal disease which would preclude the adequate oral absorption of medications.
12. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current active pneumonitis/interstitial lung disease.
13. History of current active tuberculosis.
14. Has had an allogenic tissue/solid organ transplant.
15. History of uncontrolled hypertension (≥ 180/110), dyspnoea at rest, or chronic therapy with oxygen.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.

Exclusion Criteria (Registration):

In addition to the above listed pre-registration exclusion criteria, any one of the following is regarded as a criterion for exclusion from registration to the study:

1. Have received treatment with any systemic anti-cancer therapy (including hormonal therapy), non-CNS radiation or experimental agent within 28 days of registration, except for participants with ER-positive breast cancer.
2. Have any toxicity related to prior cancer therapies that has not resolved to ≤ Grade 1, with the following exceptions:

   1. Alopecia
   2. Neuropathy, which must have resolved to ≤ Grade 2
   3. Menopausal symptoms.
3. Any untreated brain lesions > 2.0 cm in size, unless discussed with BCT and Study Chair and approval for registration is given.
4. Ongoing use of systemic corticosteroids for control of symptoms of brain metastases at a total daily dose of > 2 mg of dexamethasone (or equivalent). However, patients on a chronic stable dose of ≤ 2 mg total daily of dexamethasone (or equivalent) may be eligible with discussion and approval by BCT and the Study Chair.
5. Any brain lesion thought to require immediate local therapy, including (but not limited to) a lesion in an anatomic site where increase in size or possible treatment-related oedema may pose risk to patient (e.g. brain stem lesions). Participants who undergo local treatment for such lesions identified by screening contrast brain MRI may still be eligible for the study based on criteria described under Registration Inclusion Criteria 4.
6. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 450 ms from a single ECG.
7. Use of a strong CYP2C8 inhibitor within 5 half-lives of the inhibitor, or a strong CYP3A4 or CYP2C8 inducer within 5 days before the first dose of study treatment. Use of sensitive CYP3A substrates should be avoided 2 weeks before registration and during study treatment.
8. Treatment with botanical preparations (e.g. herbal supplements) and traditional Chinese medicines, intended for general health support or to treat the disease under study, within 7 days before registration.
9. Active infection requiring systemic therapy.
10. Administration of a live/live attenuated vaccine within 30 days before registration.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed, however intranasal influenza vaccines (e.g. FluMist®) are live attenuated vaccines and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) in the PD-L1 positive cohort | Through to study completion, an average of 24 months
  Defined as complete response (CR) or partial response (PR) assessed as per RECIST 1.1

SECONDARY OUTCOMES:
Objective response rate (ORR) in the PD-L1 negative/unknown cohort | Through to study completion, an average of 24 months
  Defined as complete response (CR) or partial response (PR) assessed as per RECIST 1.1
Progression free survival (PFS) in each PD-L1 cohort | From the time of registration until documented disease progression by RECIST 1.1 or death due to any cause (whichever occurs first), assessed up to 24 months
  Defined as the time from start of study treatment until documented disease progression by RECIST 1.1 or death due to any cause (whichever occurs first) based on local investigator assessment.
Duration of response (DoR) in each PD-L1 cohort | From the time of registration to first documentation of progressive disease or death, assessed up to 24 months
  Defined as the time from first documentation of CR or PR by RECIST 1.1 to first documentation of progressive disease or death, in the subset of participants with objective response.
Clinical benefit rate (CBR) in each PD-L1 cohort | From time of registration to CR or PR, assessed up to 24 months
  Defined as stable disease (SD) for >= 6 months after starting study treatment, or best response of CR or PR.
Overall survival (OS) in each PD-L1 cohort | From time of registration until death from any cause, assessed at 24 months
  Defined as from the time from start of study treatment to death from any cause
Incidence of treatment-emergent adverse events [Safety] | From registration until 30 days after end of study treatment
  Assessed as worst grade of adverse events (AEs) and serious adverse events (SAE) documented using NCI-CTCAE 5.0.
Incidence of treatment-emergent adverse events [Tolerability of tucatinib] | From start of study treatment to the end of study treatment, assessed at 24 months
  Assessed by tucatinib dose holding, dose reduction, drug discontinuation.
Incidence of treatment-emergent adverse events [Tolerability of pembrolizumab] | From start of study treatment to end of study treatment, assessed at 24 months
  Assessed by pembrolizumab dose holding, dose reduction, drug discontinuation.

OTHER OUTCOMES:
CNS progression in each PD-L1 cohort in participants with or without evidence of brain metastases at baseline by local image review. | From the start of study treatment to the date of first CNS progression, assessed at 24 months
  Time to CNS progression per RECIST 1.1 measured from the start of study treatment to the date of first CNS progression. Non-CNS progression and death will be considered competing events.
Extra-cranial PFS in each PD-L1 cohort | Until documented disease progression, assessed at 24 months
  PFS excluding CNS progression defined as the time from start of study treatment until documented disease progression by RECIST 1.1 or death due to any cause (whichever occurs first) based on local investigator assessment.
PFS in participants with or without evidence of brain metastases at baseline in each PD-L1 cohort | Until documented disease progression or death due to any cause, assessed at 24 months
  Defined as the time from start of study treatment until documented disease progression by RECIST 1.1 or death due to any cause (whichever occurs first) based on local investigator assessment.
Identify potential biomarkers of response - PD-L1 | At screening
  PD-L1 protein status (positive or negative) will be evaluated centrally by immunohistochemistry (IHC) using the 22C3 pharmDx PD-L1 assay. PD-L1 is positive by a MSD Combined Positive Score (CPS) of ≥ 10.
Identify potential biomarkers of response - Tumour infiltrating lymphocytes (TILs) | At baseline and 3 weeks after starting study treatment.
  Stromal Tumour Infiltrating Lymphocyte percentage (TIL%) will be recorded as per www.tilsinbreastcancer.org. Objective responses will be assessed as a function of TILs adjusted for other clinico-pathological factors, the hypothesis being that high levels of TILs will be associated with a higher rate of objective responses in this study.
Identify potential biomarkers of response - DNA and RNA | At baseline
  To understand the molecular landscape (mutations, rearrangements and copy number changes) associated with HER2-positive, PD-L1 expressing tumours as well as response or resistance to the investigational study treatment.
Identify potential biomarkers of response - ctDNA | Before first dose of study drug, before dose at Cycle 3 and Cycle 8 (each Cycle is 21 days), 30 days after stopping study treatment and/or at disease progression, assessed at 24 months
  To track and monitor tumour dynamics during treatment.
Identify potential biomarkers of response - peripheral blood mononuclear cells (PBMC) | At Baseline, every 6 weeks for 24 weeks, then every 9 weeks until disease progression, 30 days after stopping study treatment and/or at progression, assessed at 24 months
  To determine evidence of immune activation.

CONTACTS AND LOCATIONS:
Overall Officials: Heath Badger, Study Director — Breast Cancer Trials, Australia and New Zealand; Sherene Loi, Prof, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (15):
- Australia (15):
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Nepean Cancer Care Centre, Kingswood, New South Wales
  - Macquarie University, Macquarie Park, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Icon Cancer Centre Hobart, Hobart, Tasmania
  - Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Parkville, Victoria
  - Epworth Richmond Hospital, Richmond, Victoria
  - Sunshine Hospital, St Albans, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Refer to BCT Data Sharing Guidelines (contact concept@bctrials.org.au for further details).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available for request after publication of the main/final study results; no end date. Note that there may be additional circumstances preventing BCT from sharing requested data as outlined in the BCT Data Sharing Guidelines.
Access Criteria: Researchers need to submit a research proposal (concept@bctrials.org.au) and BCT Data Request Application, which is then assessed by BCT as having appropriate scientific value.

REFERENCES:
- See also: Breast Cancer Trials, Australia and New Zealand — http://www.breastcancertrials.org.au